CLINICAL TRIAL: NCT03108807
Title: Combined Use of the National Early Warning Score and D-dimer to Identify Medical Patients At Low Risk of 30-day Mortality in a Danish Emergency Department
Brief Title: National Early Warning Score and D-dimer to Identify Medical Patients At Low Risk of 30-day Mortality
Status: Completed | Type: Observational
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Mikkel Brabrand, MD, PhD, clinical associate professor, Esbjerg Hospital - University Hospital of Southern Denmark
Other Study IDs: S-20170005
Record Dates: First submitted 2017-04-03; First posted 2017-04-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Medical Patients in the Emergency Department
Keywords: Emergency Department; Medical patients; D-dimer; National Early Warning Score; NEWS; 30-days mortality; Mortality
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: D-dimer test — D-dimer test

SUMMARY:
The aim is to determine if the National Early Warning Score combined with plasma D-dimer levels can be used in risk stratification of acutely ill medical patients presenting to a Danish Emergency Department. The investigators wish to identify patients at low risk of mortality within 30 days.

DETAILED DESCRIPTION:
Large increases in emergency admissions are raising concerns about whether all admissions are necessary. If there was a fast and reliable system that could be used to determine the risk of all medical patients, many low-risk patients could be safely returned to primary care or outpatient follow-up clinics.

The investigators wish to determine, if the combination of the National Early Warning Score and plasma D-dimer levels can be used to identify patients at low risk of mortality within 30 days in an unselected group of medical patients presenting to a Danish Emergency Department.

This is a prospective observational study that will be performed on adult medical patients referred to the Emergency Department of a Danish hospital to be assessed for possible admission. The study will be performed in the Emergency Department of Hospital of South West Jutland in the region of Southern Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Emergency Department of Hospital of South West Jutland
* Requirement of any blood test
* Age 18 years
* Informed consent given

Exclusion Criteria:

* Age 18 years
* Informed consent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An unselected group of consecutive patients in a Danish Emergency Department.
Sampling Method: Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-08-19 (Actual); Study Completion 2017-08-19 (Actual)

PRIMARY OUTCOMES:
30-days mortality | 30 days
  mortality within 30 days after assessment will be determined for all patients using data extracted from the Danish Civil Registration System patients using data extracted from the Danish Civil Registration System

SECONDARY OUTCOMES:
Hospital length of stay (LOS) | 30 days
  length of stay will be calculated from the time of the patients' arrival at the hospital to the moment of the discharge for all patients using data extracted from the Danish National Patient Registry
Readmissions within 30 days | 30 days
  readmissions within 30 days after primary assessment will be determined for all patients using data extracted from the Danish National Patient Registry

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Brabrand, MD, PhD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (1):
- Hospital of South West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nickel CH, Kuster T, Keil C, Messmer AS, Geigy N, Bingisser R. Risk stratification using D-dimers in patients presenting to the emergency department with nonspecific complaints. Eur J Intern Med. 2016 Jun;31:20-4. doi: 10.1016/j.ejim.2016.03.006. Epub 2016 Apr 1. PMID 27053291
- [Background] Nickel CH, Kellett J, Cooksley T, Bingisser R, Henriksen DP, Brabrand M. Combined use of the National Early Warning Score and D-dimer levels to predict 30-day and 365-day mortality in medical patients. Resuscitation. 2016 Sep;106:49-52. doi: 10.1016/j.resuscitation.2016.06.012. Epub 2016 Jun 20. PMID 27339095
- [Derived] Nickel CH, Kellett J, Nieves Ortega R, Lyngholm L, Wasingya-Kasereka L, Brabrand M. Mobility Identifies Acutely Ill Patients at Low Risk of In-Hospital Mortality: A Prospective Multicenter Study. Chest. 2019 Aug;156(2):316-322. doi: 10.1016/j.chest.2019.04.001. Epub 2019 Apr 11. PMID 30981722